CLINICAL TRIAL: NCT05849506
Title: Touch on One Thumb, RSI on the Other Thumb: Which Surgery Shows Better Results: An Ambidirectional Trial
Brief Title: Touch on One Thumb, RSI on the Other Thumb: Which Surgery Shows Better Results
Status: Completed | Type: Observational
Sponsor: Schulthess Klinik (Other)
Responsible Party: Sponsor
Other Study IDs: OE-0203
Record Dates: First submitted 2023-03-30; First posted 2023-05-09 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Osteoarthritis Thumb; Joint Diseases; Musculoskeletal Diseases or Conditions; Osteoarthritis; Arthrosis of First Carpometacarpal Joint
Keywords: Touch® prothesis; RSI; Resection-suspension-interposition arthroplasty; Thumb carpometacarpal joint; Dual mobility prosthesis
MeSH Terms: conditions — Joint Diseases; Musculoskeletal Diseases; Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Touch-RSI: The group consists of patients with a Touch® implant in one thumb and an RSI arthroplasty in the other thumb.
  Intervention: Patient questionnaire and clinical examination to investigate differences between the thumb with a Touch® implant and the thumb with an RSI.
  Interventions: Device: Touch® Prosthesis

INTERVENTIONS:
Device: Touch® Prosthesis — The Touch® prosthesis is a medical device approved in Switzerland, which is an effective surgical treatment for advanced CMC I osteoarthritis.

SUMMARY:
The study aims to determine whether CMC I arthroplasty using a Touch® implant results in higher patient satisfaction compared to RSI arthroplasty in the medium-term in patients with primary thumb osteoarthritis. Additionally, the study compares the patients' clinical and self-reported outcomes between the Touch® implant and the RSI arthroplasty. Therefore, patients with a Touch® implant in one thumb and an RSI arthroplasty in the other thumb will be recruited.

DETAILED DESCRIPTION:
Patients suffering from osteoarthritis in the first carpometacarpal joint (CMC I OA) are often surgically treated with a resection-suspension-interposition (RSI) arthroplasty. An alternative technique is an arthroplasty with a Touch® implant. There is a growing body of evidence indicating that patients with a Touch® prosthesis recover significantly faster and return to work more quickly than patients after an RSI arthroplasty. However, there have been no studies comparing the two operations in the same patient. By recruiting patients with a Touch® implant in one thumb and an RSI arthroplasty in the other thumb, this study aims to investigate whether CMC I arthroplasty using a Touch® implant leads to higher patient satisfaction compared to RSI arthroplasty in the medium-term. Further patient-reported and clinical outcomes will be assessed to compare the two surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent signed by the patient.
* Patient is diagnosed with primary OA in both CMC I joints and was operated with a Touch® prosthesis on one thumb and with an RSI arthroplasty on the other thumb.

Exclusion Criteria:

* Patient with any type of revision surgery at the CMC I joint
* Patient underwent hand surgery within the last three months
* Legal incompetence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients with CMC I joint osteoarthritis. They have a Touch® prosthesis in one thumb and an RSI arthroplasty in the other.
Sampling Method: Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2023-06-21 (Actual); Primary Completion 2024-02-10 (Actual); Study Completion 2024-02-10 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction wiht treatment result using 5-point Likert scale | Follow-up at least 3 months to 12 years after surgery
  5-point Likert scale ranging from 1 (very dissatisfied) to 5 (very satisfied)

SECONDARY OUTCOMES:
Sociodemographic information | Follow-up at least 3 months to 12 years after surgery
  Questionnaire
Additional aspects of patient satisfaction with treatment | Follow-up at least 3 months to 12 years after surgery
  Questionnaire
Differences between both thumbs | Follow-up at least 3 months to 12 years after surgery
  Questionnaire
Brief Michigan Hand Outcomes Questionnaire (MHQ) | Follow-up at least 3 months to 12 years after surgery
  The german version of the brief MHQ will be used to assess patient-reported hand function. The score ranges from 0 to 100 with higher scores indicating better hand function.
Grip strength assessed with Jamar Dynamometer | Follow-up at least 3 months to 12 years after surgery
  Jamar Dynamometer
Key pinch strength assessed with pinch gauge | Follow-up at least 3 months to 12 years after surgery
  Pinch gauge
Range of motion of the humb metacarpal (MCP) and interphalangeal (IP) joint assessed with a goniometer | Follow-up at least 3 months to 12 years after surgery
  Used to measure flexion and extension of the thumb metacarpal (MCP) and interphalangeal (IP) joint. The evaluation of active thumb opposition is based on the Kapandji index, ranging from 1 (can touch only the lateral side of the index finger) to 10 (can reach the volar crease of the hand).
Pain at rest and during activities of daily living (ADL) assessed using Numeric rating scales (NRS) | Follow-up at least 3 months to 12 years after surgery
  NRS ranging from 0 (no pain) to 10 (worst pain)
Radiographs of both thumbs | Follow-up at least 3 months to 12 years after surgery
  To monitor the implant and to assess the scaphometacarpal distance, which can be used to identify migration of the thumb metacarpal bone, a phenomenon often observed after trapeziectomy.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel B. Herren, Dr. med., Principal Investigator — Schulthess Klinik
Locations (1):
- Schulthess Klinik, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No